CLINICAL TRIAL: NCT04626882
Title: OPtimal TIming of Fractional Flow Reserve-Guided Complete RevascularizatiON for Non-Infarct Related Artery in ST-Segment Elevation Myocardial Infarction With Multivessel Disease (OPTION-STEMI)
Brief Title: Timing of FFR-guided PCI for Non-IRA in STEMI and MVD (OPTION-STEMI)
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Chonnam National University Hospital (Other)
Responsible Party: Principal Investigator, Min Chul Kim, Associate Professor, Chonnam National University Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CNUH-2019-318
Record Dates: First submitted 2020-11-02; First posted 2020-11-13 (Actual); Last update posted 2025-05-30 (Actual); Status verified 2025-05

CONDITIONS: Myocardial Infarction, Acute; Multi-Vessel Coronary Artery Stenosis
MeSH Terms: conditions — Myocardial Infarction

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Staged in-hospital CR (complete revascularization) (Active Comparator): Non-infarct related artery (IRA) will be revascularized in other day (during hospitalization) after PCI for IRA. Non-IRA lesion which have equal or more than 70% diameter stenosis by visual estimation will be revascularized without FFR evaluation. Non-IRA lesion with diameter stenosis 50-70% by visual estimation will be evaluated using FFR device. In case of FFR value more than 0.8, non-IRA lesion wll be deferred without PCI. If FFR value was equal or less than 0.8, non-IRA lesion will be revascularized.
  Interventions: Procedure: Staged in-hospital or Immediate complete revascularization
- Immediate CR (complete revascularization) (Experimental): Non-infarct related artery (IRA) will be revascularized immediately after PCI for IRA (during primary PCI). Non-IRA lesion which have equal or more than 70% diameter stenosis by visual estimation will be revascularized without FFR evaluation. Non-IRA lesion with diameter stenosis 50-70% by visual estimation will be evaluated using FFR device. In case of FFR value more than 0.8, non-IRA lesion wll be deferred without PCI. If FFR value was equal or less than 0.8, non-IRA lesion will be revascularized.
  Interventions: Procedure: Staged in-hospital or Immediate complete revascularization

INTERVENTIONS:
Procedure: Staged in-hospital or Immediate complete revascularization — Patients with ST-segment elevation myocardial infarction and multivessel disease will be randomized after primary PCI for IRA. All patients will be randomized to immediate complete revascularization group or staged revascularization group by 1:1 fashion. Non-IRA lesion which have equal or more than 70% diameter stenosis by visual estimation will be revascularized without FFR evaluation. Non-IRA lesion with diameter stenosis 50-70% by visual estimation will be evaluated using FFR device. In case of FFR value more than 0.8, non-IRA lesion wll be deferred without PCI. If FFR value was equal or less than 0.8, non-IRA lesion will be revascularized.

SUMMARY:
Patients with STEMI (ST-segment elevation myocardial infarction) with multivessel disease which have PCI (percutaneous coronary intervention)-suitable non-IRA (infarct related artery) will be randomized to immediate complete revascularization group or staged revascularization group by 1:1 fashion. Non-IRA lesion which have equal or more than 70% diameter stenosis by visual estimation will be revascularized without FFR (fractional flow reserve) evaluation. Non-IRA lesion with diameter stenosis 50-70% by visual estimation will be evaluated using FFR device. In case of FFR value more than 0.8, non-IRA lesion wll be deferred without PCI. If FFR value was equal or less than 0.8, non-IRA lesion will be revascularized.

DETAILED DESCRIPTION:
Study objectives:

To determine the optimal timing of non-infarct related artery (IRA) percutaneous coronary intervention (PCI) with the aid of FFR (fractional flow reserve) (immediate complete revascularization during primary angioplasty vs. staged procedure for non-IRA PCI) in patients with ST-segment elevation myocardial infarction with multivessel disease (MVD).

Study hypothesis:

Complete revascularization (CR) at index procedure is not inferior to staged in-hospital CR in patients with STEMI and MVD who undergoing FFR-guided revascularization for non-IRA.

Background:

Multivessel coronary artery disease (MVD) is a common clinical condition, about 40-65% of all primary angioplasty, encountered by interventional cardiologists in ST-segment elevation myocardial infarction (STEMI), and it is associated with poorer clinical outcomes than single-vessel disease. Older guidelines recommended culprit-vessel only revascularization (CVR) during primary angioplasty, except in patient that are hemodynamically unstable. Several recent studies have reported improved clinical outcomes in these patients with multivessel percutaneous coronary intervention (PCI), and others reported promising results from CVR followed by elective second-stage PCI at non-infarct related artery (non-IRA) with significant stenosis. However, there has been no consensus of optimal revascularization strategy in this circumstance.

Recently, several large-scaled randomized controlled trials were conducted about this issue, and confirmed the benefit of immediate complete revascularization during primary angioplasty compared to CVR. Furthermore, fractional flow reserve (FFR)-guided PCI at non-IRA was more effective than angiography-guided PCI at non-IRA for reducing repeat revascularization by either immediate multivessel PCI strategy or staged PCI strategy in the other trials.

Although FFR is a well-known tool to evaluate significant ischemia of moderate stenosis, the most studies regarding FFR enrolled patients without acute myocardial infarction (AMI). Timing of non-IRA PCI is also uncertain. After promising results of above-mentioned randomized trials, current guideline recommendation of multivessel PCI (immediate or staged) was upgraded. However, current guidelines simply mentioned about the timing of non-IRA PCI which recommends complete revascularization during initial hospitalization by either of immediate of staged PCI strategy.

Therefore, the investigators planned to perform prospective, open-label, multicenter, non-inferiority trial to evaluate the efficacy and safety of immediate complete revascularization (PCI for both IRA and non-IRA during primary angioplasty) compared to staged PCI strategy of non-IRA (primary angioplasty for IRA followed by non-IRA PCI after several days). PCI procedure at non-IRA with diameter stenosis between 50 and 70% should be conducted with the aid of FFR, and non-IRA with diameter stenosis ≥ 70% will be revascularized without FFR.

Study procedure:

Patients will be randomized after primary PCI for IRA. Non-IRA lesion which have equal or more than 70% diameter stenosis by visual estimation will be revascularized without FFR evaluation. Non-IRA lesion with diameter stenosis 50-70% by visual estimation will be evaluated using FFR device. In case of FFR value more than 0.8, non-IRA lesion wll be deferred without PCI. If FFR value was equal or less than 0.8, non-IRA lesion will be revascularized.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 19 years old
* ST-segment elevation myocardial infarction

  * ST-segment elevation in at least 2 contiguous leads or,
  * New onset left bundle branch block
* Primary PCI within 12 hours after symptom development
* Multivessel disease: Non-IRA with at least 2.5 mm diameter and 50% diameter stenosis by visual estimation
* Patient's or protector's agreement about study design and the risk of PCI

Exclusion Criteria:

* Cardiogenic shock at initial presentation or after treatment of IRA
* Unprotected left main coronary artery disease with at least 50% diameter stenosis by visual estimation
* TIMI (Thrombolysis in Myocardial Infarction) flow at non-IRA ≤ 2
* Severe procedural complications (e.g. persistent no-reflow phenomenon, coronary artery perforation) which restricts study enrollment by operators' decision
* Non-IRA lesion not suitable for PCI treatment by operators' decision
* Chronic total occlusion at non-IRA
* History of anaphylaxis to contrast agent
* Pregnancy and lactation
* Life expectancy < 1-year
* Severe valvular disease
* History of CABG (coronary artery bypass graft), or planned CABG
* Fibrinolysis before admission
* Severe asthma
* Patient's refusal to participate in study

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 994 (Actual)
Dates: Start 2019-12-30 (Actual); Primary Completion 2025-01-15 (Actual); Study Completion 2029-12-31 (Estimated)

PRIMARY OUTCOMES:
Cumulative incidence rate of all-cause death, non-fatal myocardial infarction, or all unplanned revascularization at 1 year from baseline | Index admission to 12 months
  Composite endpoint of all-cause death, non-fatal myocardial infarction, or all unplanned revascularization at 1 year after index percutaneous coronary intervention

SECONDARY OUTCOMES:
Rate of contrast-induced nephropathy during index admission | During index admission
  Rate of contrast-induced nephropathy during index admission
Cumulative incidence rate of all unplanned revascularization at each visit | Index admission, 1 month, 6 months, 12 months, 24 months, 36 months, 48 months, 60 months
  Cumulative incidence rate of all unplanned revascularization at each visit
Cumulative incidence rate of target-lesion revascularization at each visit | Index admission, 1 month, 6 months, 12 months, 24 months, 36 months, 48 months, 60 months
  Cumulative incidence rate of target-lesion revascularization at each visit
Cumulative incidence rate of target-vessel revascularization at each visit | Index admission, 1 month, 6 months, 12 months, 24 months, 36 months, 48 months, 60 months
  Cumulative incidence rate of target-vessel revascularization at each visit
Cumulative incidence rate of non-target vessel revascularization at each visit | Index admission, 1 month, 6 months, 12 months, 24 months, 36 months, 48 months, 60 months
  Cumulative incidence rate of non-target vessel revascularization at each visit
Cumulative incidence rate of all-cause death at each visit | Index admission, 1 month, 6 months, 12 months, 24 months, 36 months, 48 months, 60 months
  Cumulative incidence rate of all-cause death at each visit
Cumulative incidence rate of cardiac death at each visit | Index admission, 1 month, 6 months, 12 months, 24 months, 36 months, 48 months, 60 months
  Cumulative incidence rate of cardiac death at each visit
Cumulative incidence rate of non-cardiac death at each visit | Index admission, 1 month, 6 months, 12 months, 24 months, 36 months, 48 months, 60 months
  Cumulative incidence rate of non-cardiac death at each visit
Cumulative incidence rate of non-fatal myocardial infarction at each visit | Index admission, 1 month, 6 months, 12 months, 24 months, 36 months, 48 months, 60 months
  Cumulative incidence rate of non-fatal myocardial infarction at each visit
Cumulative incidence rate of hospitalization for unstable angina at each visit | Index admission, 1 month, 6 months, 12 months, 24 months, 36 months, 48 months, 60 months
  Cumulative incidence rate of hospitalization for unstable angina at each visit
Cumulative incidence rate of hospitalization for heart failure at each visit | Index admission, 1 month, 6 months, 12 months, 24 months, 36 months, 48 months, 60 months
  Cumulative incidence rate of hospitalization for heart failure at each visit
Cumulative incidence rate of definite or probable stent thrombosis at each visit | Index admission, 1 month, 6 months, 12 months, 24 months, 36 months, 48 months, 60 months
  Cumulative incidence rate of definite or probable stent thrombosis at each visit
Cumulative incidence rate of ischemic and hemorrhagic stroke at each visit | Index admission, 1 month, 6 months, 12 months, 24 months, 36 months, 48 months, 60 months
  Cumulative incidence rate of ischemic and hemorrhagic stroke at each visit
Cumulative incidence rate of major bleeding (BARC definitions type 3 or 5) at each visit | Index admission, 1 month, 6 months, 12 months, 24 months, 36 months, 48 months, 60 months
  Cumulative incidence rate of major bleeding (BARC definitions type 3 or 5) at each visit
Cumulative incidence rate of all-cause death, non-fatal myocardial infarction, or all unplanned revascularization at 1 year from baseline | Index admission, 1 month, 6 months, 12 months, 24 months, 36 months, 48 months, 60 months
  Composite endpoint of all-cause death, non-fatal myocardial infarction, or all unplanned revascularization at 1 year after index percutaneous coronary intervention

CONTACTS AND LOCATIONS:
Overall Officials: Youngkeun Ahn, MD, Principal Investigator — Chonnam National University Hospital
Locations (14):
- South Korea (14):
  - The Catholic University of Korea, Bucheon St. Mary's Hospital, Bucheon-si
  - Gyeongsang National University Changwon Hospital, Changwon
  - Yeongnam University Medical Center, Daegu
  - GangNeung Asan Hospital, Gangneung
  - Chonnam National University Hospital, Gwangju
  - Chonbuk National University Hospital, Jeonju
  - Presbyterian Medical Center, Jeonju
  - Gyeongsang National University Hospital, Jinju
  - Koera University Guro Hospital, Seoul
  - Kyung Hee University Hospital, Seoul
  - The Catholic University of Korea, Seoul St. Mary's Hospital, Seoul
  - St. Carollo General Hospital, Suncheon
  - The Catholic University of Korea, Uijeongbu St. Mary's Hospital, Uijeongbu-si
  - Yonsei University, Wonju Severance Christian Hospital, Wŏnju

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Kim MC, Ahn JH, Hyun DY, Lim Y, Cho KH, Lee SH, Park S, Oh S, Sim DS, Hong YJ, Kim JH, Jeong MH, Cho JH, Lee SR, Kang DO, Hwang JY, Youn YJ, Lee JH, Jeong YH, Ahn JH, Kim DB, Choo EH, Kim CJ, Kim W, Rhew JY, Park JI, Yoo SY, Ahn Y; OPTION-STEMI Investigators. Immediate versus staged complete revascularisation during index admission in patients with ST-segment elevation myocardial infarction and multivessel disease (OPTION-STEMI): a multicentre, non-inferiority, open-label, randomised trial. Lancet. 2025 Sep 6;406(10507):1032-1043. doi: 10.1016/S0140-6736(25)01529-6. Epub 2025 Aug 31. PMID 40902612
- [Derived] Kim MC, Ahn JH, Hyun DY, Lim Y, Lee SH, Oh S, Cho KH, Sim DS, Hong YJ, Kim JH, Jeong MH, Cho JH, Lee SR, Kang DO, Hwang JY, Youn YJ, Jeong YH, Park Y, Kim DB, Choo EH, Kim CJ, Kim W, Rhew JY, Lee JH, Yoo SY, Ahn Y; OPTION-STEMI Investigators. Timing of fractional flow reserve-guided complete revascularization in patients with ST-segment elevation myocardial infarction with multivessel disease: Rationale and design of the OPTION-STEMI trial. Am Heart J. 2024 Jul;273:35-43. doi: 10.1016/j.ahj.2024.03.017. Epub 2024 Apr 18. PMID 38641031